CLINICAL TRIAL: NCT06159335
Title: Use of 18F-Fluciclovine PET for Discerning Tumor From Treatment Change in Patients With Brain Metastases Undergoing Immunotherapy
Brief Title: 18F-FLUC PET/MR in Patients With Brain Mets
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Blue Earth Diagnostics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-1082; NCI-2024-06018 (Registry Identifier: NCI Trial ID); Protocol Version 11/20/2025 (Other: UW Madison); A539300 (Other: UW Madison); UW23061 (Other: UW Madison)
Record Dates: First submitted 2023-11-28; First posted 2023-12-06 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-02

CONDITIONS: Brain Metastasis; Radiation Therapy; Immunotherapy, Active
MeSH Terms: conditions — Brain Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- PET-MRI (Experimental): Participants will undergo F-Fluciclovine PET radiotracer and MRI
  Interventions: Radiation: F-Fluciclovine radiotracer

INTERVENTIONS:
Radiation: F-Fluciclovine radiotracer — Participants will receive PET radiotracer and MRI

SUMMARY:
The goal of this clinical trial is to use new imaging methods to help in finding out whether the imaging shows that there is a tumor in people with a brain metastasis. The main question it aims to answer is whether positron emission tomography (PET) and magnetic resonance imaging (MRI) find cancerous tissue better than other types of imagining.

Participants will undergo a single PET/MRI scan, followed by a separate MRI scan with a tracer. Study participation will last about 3 hours.

DETAILED DESCRIPTION:
The purpose of this research is to utilize new imaging methods to aid in assessing whether imaging shows presence of tumor. Developing imaging technologies is critical for more accurately identifying location and amount of tumor, which will then lead to improvements in future cancer therapy.

This study aims to evaluate imaging methods known as PET and MRI to improve detection of cancerous tissue better than the types of imaging that are currently available.

These methods are conducted on the same machine as conventional MRI that uses a powerful magnet, radio waves, and a computer to create detailed images. Both the PET and MRI methods look at the number of proteins a tumor has. The more proteins, the more likely there is tumor relative to normal brain tissue.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able and willing to provide informed consent
* Has a brain metastasis diagnosis with at least one single visible contrast enhancing metastatic lesion on brain MRI
* Received radiation therapy at some point in the last 2 years
* Is currently being treated with or has been treated with any other concurrent systemic therapy (multi-modal therapy) in the past 6 months, which would include immunotherapy, targeted therapy, or systemic chemotherapy, immunotherapy, or chemotherapy following radiation therapy.
* Patients are eligible for the study if their most recent standard-of-care MRI, used to assess disease location and extent, raises the question of tumor recurrence versus treatment-related changes. This concern can be noted by the radiologist or other members of the multidisciplinary care team, such as during a multidisciplinary conference. Additionally, if there are clinical concerns based on evolving exam findings or symptoms, and the treating physician suspects progression versus treatment-induced changes, the patient is also eligible for the study.
* Be able to lie still for 30-60 minutes during the imaging procedure
* Willing and able to undergo PET/MRI or PET/CT
* Patients requiring intravenous (IV) conscious sedation for imaging are not eligible; patients requiring mild, oral anxiolytics for the clinical MRI will be allowed to participate as long as the following criteria are met:

  * The subject has their own prescription for the medication
  * The informed consent process is conducted prior to the self-administration of this medication
  * They come to the research visit with a driver

Exclusion Criteria:

* Subject unable or unwilling to provide informed consent
* Subject is pregnant
* Subject with contraindication(s) to or inability to undergo a PET/MR or PET/CT
* Known allergy to 18F-Fluciclovine or any of its excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-01-10 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Amino acid uptake into tumor tissue | 3 hours
  Using 18F-Fluciclovine PET, compare amino acid uptake into brain tumor tissue with uptake in normal brain tissue. Higher uptake is hypothesized to indicate malignancy

CONTACTS AND LOCATIONS:
Overall Officials: Michael Veronesi, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No